CLINICAL TRIAL: NCT01982240
Title: A Randomized, 12-Week, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Plecanatide (3.0 and 6.0 mg) in Patients With Chronic Idiopathic Constipation (The CIC3 Study)
Brief Title: 12-Week Study of Plecanatide for CIC (The CIC3 Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP304203-00
Record Dates: First submitted 2013-11-05; First posted 2013-11-13 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Chronic Idiopathic Constipation
Keywords: CIC; Constipation; Chronic Constipation; Synergy; Plecanatide
MeSH Terms: conditions — Constipation | interventions — plecanatide; Bisacodyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Plecanatide 3.0 mg (Active Comparator): Plecanatide tablets 3.0 mg QD for 12 weeks
  Interventions: Drug: Plecanatide
- Plecanatide 6.0 mg (Active Comparator): Plecanatide tablets 6.0 mg QD for 12 weeks
  Interventions: Drug: Plecanatide
- Placebo (Placebo Comparator): Matching placebo tablets QD for 12 weeks
  Interventions: Drug: Placebo
- Bisacodyl (Other): Rescue medication
  Interventions: Drug: Bisacodyl

INTERVENTIONS:
Drug: Plecanatide — Plecanatide tablets QD for 12 weeks
  Other Names: Trulance
  Arms: Plecanatide 3.0 mg; Plecanatide 6.0 mg
Drug: Placebo — Matching placebo tablets QD for 12 weeks
  Other Names: Trulance placebo
  Arms: Placebo
Drug: Bisacodyl — Rescue medication
  Other Names: Dulcolax
  Arms: Bisacodyl

SUMMARY:
The purpose of this study is to confirm that the investigational medication, plecanatide, is safe and effective in treating chronic idiopathic constipation.

DETAILED DESCRIPTION:
This is a randomized, 12-week, double-blind, placebo-controlled, study in approximately 1350 adult male and female patients with CIC comparing 2 doses of plecanatide to placebo. The study will be conducted at approximately 180 clinical study sites in the United States (US) and Canada. The primary objective of the study is to evaluate the efficacy and safety of 3.0 and 6.0 mg of plecanatide administered once daily (QD) for 12 weeks in a population of patients with CIC. The study population will include only patients without other causes of constipation or other chronic conditions that could interfere with study assessments. Patients may not take laxatives (with the exception of the study-provided rescue medication, bisacodyl 5mg tablets), or a number of prohibited drugs that are known to cause constipation or diarrhea, during study participation.

There are 6 scheduled study visits, including the screening and follow-up visits. The planned duration of participation in this study will be 112 days and up to 155 days, with washout and all visit windows considered.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-80, inclusive
* Meets modified Rome III criteria for functional chronic idiopathic constipation for at least 3 months with symptom onset for at least 6 months
* Completed a colonoscopy in accordance with AGA colon cancer screening guidelines (5 years), with no clinically significant findings
* Willing to maintain a stable diet during the study

Exclusion Criteria:

* Loose stool (mushy) or watery (Bristol score 6 or 7) stool in the absence of any laxative or prohibited medicine for > 25% of BMs during the 3 months prior to screening visit OR during the 14 day pre-treatment assessment
* Active peptic ulcer disease, diabetes or hypertension not adequately treated or not stable
* History of cathartic colon, laxative, enema abuse, or ischemic colitis
* Fecal impaction within 3 months of screening
* Patient has had /has any: diseases or conditions associated with constipation (GI or CNS), structural abnormality of the GI tract or gastric bypass surgery, pelvic floor dysfunction, pseudo-obstruction, active infectious gastritis, diverticulitis, anal fissures or any disease or condition that can affect GI motility or defecation or can be associated with abdominal pain
* Unexplained and clinically significant "alarm symptoms" including lower GI bleeding, iron-deficiency anemia, weight loss or systemic signs of infection or colitis
* Major surgery, stroke or MI within 60 days of screening
* Participated in a previous plecanatide clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1394 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Layton, Study Director — Synergy Pharmaceuticals Inc.
Locations (157):
- United States (146):
  - Synergy Research Site, Birmingham, Alabama
  - Synergy Research Site, Dothan, Alabama
  - Synergy Research Site, Gulf Shores, Alabama
  - Synergy Research Site, Huntsville, Alabama
  - Synergy Research Site, Mobile, Alabama
  - Synergy Research Site, Mesa, Arizona
  - Synergy Research Site, Phoenix, Arizona
  - Synergy Research Site, Tempe, Arizona
  - Synergy Research Site, Tucson, Arizona
  - Synergy Research Site, Hot Springs, Arkansas
  - Synergy Research Site, Little Rock, Arkansas
  - Synergy Research Site, North Little Rock, Arkansas
  - Synergy Research Site, Anaheim, California
  - Synergy Research Site, Carlsbad, California
  - Synergy Research Site, Cerritos, California
  - Synergy Research Site, Chula Vista, California
  - Synergy Research Site, El Cajon, California
  - Synergy Research Site, Encinitas, California
  - Synergy Research Site, Encino, California
  - Synergy Research Site, Fountain Valley, California
  - Synergy Research Site, Fresno, California
  - Synergy Research Site, Hawaiian Gardens, California
  - Synergy Research Site, Lancaster, California
  - Synergy Research Site, Long Beach, California
  - Synergy Research Site, Los Angeles, California
  - Synergy Research Site, Mission Hills, California
  - Synergy Research Site, Murrieta, California
  - Synergy Research Site, North Hollywood, California
  - Synergy Research Site, Oceanside, California
  - Synergy Research Site, Oxnard, California
  - Synergy Research Site, Pasadena, California
  - Synergy Research Site, Poway, California
  - Synergy Research Site, Sacramento, California
  - Synergy Research Site, San Diego, California
  - Synergy Research Site, Thousand Oaks, California
  - Synergy Research Site, Colorado Springs, Colorado
  - Synergy Research Site, Denver, Colorado
  - Synergy Research Site, Littleton, Colorado
  - Synergy Research Site, Bristol, Connecticut
  - Synergy Research Site, Danbury, Connecticut
  - Synergy Research Site, Waterbury, Connecticut
  - Synergy Research Site, Boynton Beach, Florida
  - Synergy Research Site, Clearwater, Florida
  - Synergy Research Site, DeLand, Florida
  - Synergy Research Site, Fort Lauderdale, Florida
  - Synergy Research Site, Hialeah, Florida
  - Synergy Research Site, Jupiter, Florida
  - Synergy Research Site, Lakeland, Florida
  - Synergy Research Site, Lynn Haven, Florida
  - Synergy Research Site, Miami, Florida
  - Synergy Research Site, Orlando, Florida
  - Synergy Research Site, Port Orange, Florida
  - Synergy Research Site, Tampa, Florida
  - Synergy Research Site, Athens, Georgia
  - Synergy Research Site, Augusta, Georgia
  - Synergy Research Site, Decatur, Georgia
  - Synergy Research Site, Johns Creek, Georgia
  - Synergy Research Site, Oakwood, Georgia
  - Synergy Research Site, Savannah, Georgia
  - Synergy Research Site, Smyrna, Georgia
  - Synergy Research Site, Evanston, Illinois
  - Synergy Research Site, Clive, Iowa
  - Synergy Research Site, Augusta, Kansas
  - Synergy Research Site, Newton, Kansas
  - Synergy Research Site, Shawnee Mission, Kansas
  - Synergy Research Site, Wichita, Kansas
  - Synergy Research Site, Lexington, Kentucky
  - Synergy Research Site, Bastrop, Louisiana
  - Synergy Research Site, Marrero, Louisiana
  - Synergy Research Site, Metairie, Louisiana
  - Synergy Research Site, New Orleans, Louisiana
  - Synergy Research Site, Shreveport, Louisiana
  - Synergy Research Site, Chevy Chase, Maryland
  - Synergy Research Site, Boston, Massachusetts
  - Synergy Research Site, Brockton, Massachusetts
  - Synergy Research Site, New Bedford, Massachusetts
  - Synergy Research Site, Chesterfield, Michigan
  - Synergy Research Site, Flint, Michigan
  - Synergy Research Site, Rochester, Michigan
  - Synergy Research Site, Saginaw, Michigan
  - Synergy Research Site, Southfield, Michigan
  - Synergy Research Site, Biloxi, Mississippi
  - Synergy Research Site, Jackson, Mississippi
  - Synergy Research Site, St Louis, Missouri
  - Synergy Research Site, Omaha, Nebraska
  - Synergy Research Site, Henderson, Nevada
  - Synergy Research Site, Las Vegas, Nevada
  - Synergy Research Site, Reno, Nevada
  - Synergy Research Site, Lebanon, New Hampshire
  - Synergy Research Site, Lodi, New Jersey
  - Synergy Research Site, Ocean City, New Jersey
  - Synergy Research Site, Albuquerque, New Mexico
  - Synergy Research Site, Brooklyn, New York
  - Synergy Research Site, Great Neck, New York
  - Synergy Research Site, North Massapequa, New York
  - Synergy Research Site, Cary, North Carolina
  - Synergy Research Site, Chapel Hill, North Carolina
  - Synergy Research Site, Charlotte, North Carolina
  - Synergy Research Site, Greensboro, North Carolina
  - Synergy Research Site, Kinston, North Carolina
  - Synergy Research Site, Raleigh, North Carolina
  - Synergy Research Site, Wilmington, North Carolina
  - Synergy Research Site, Winston-Salem, North Carolina
  - Synergy Research Site, Fargo, North Dakota
  - Synergy Research Site, Beavercreek, Ohio
  - Synergy Research Site, Centerville, Ohio
  - Synergy Research Site, Cincinnati, Ohio
  - Synergy Research Site, Hilliard, Ohio
  - Synergy Research Site, Huber Heights, Ohio
  - Synergy Research Site, Maumee, Ohio
  - Synergy Research Site, Mentor, Ohio
  - Synergy Research Site, Oakwood, Ohio
  - Synergy Research Site, Stow, Ohio
  - Synergy Research Site, Norman, Oklahoma
  - Synergy Research Site, Oklahoma City, Oklahoma
  - Synergy Research Site, Limerick, Pennsylvania
  - Synergy Research Site, Philadelphia, Pennsylvania
  - Synergy Research Site, Smithfield, Pennsylvania
  - Synergy Research Site, Yardley, Pennsylvania
  - Synergy Research Site, Anderson, South Carolina
  - Synergy Research Site, Charleston, South Carolina
  - Synergy Research Site, Columbia, South Carolina
  - Synergy Research Site, Chattanooga, Tennessee
  - Synergy Research Site, Jackson, Tennessee
  - Synergy Research Site, Nashville, Tennessee
  - Synergy Research Site, New Tazewell, Tennessee
  - Synergy Research Site, Austin, Texas
  - Synergy Research Site, Dallas, Texas
  - Synergy Research Site, Houston, Texas
  - Synergy Research Site, Killeen, Texas
  - Synergy Research Site, Plano, Texas
  - Synergy Research Site, San Angelo, Texas
  - Synergy Research Site, San Antonio, Texas
  - Synergy Research Site, Sugar Land, Texas
  - Synergy Research Site, Logan, Utah
  - Synergy Research Site, Salt Lake City, Utah
  - Synergy Research Site, St. George, Utah
  - Synergy Research Site, Christiansburg, Virginia
  - Synergy Research Site, Henrico, Virginia
  - Synergy Research Site, Lynchburg, Virginia
  - Synergy Research Site, Norfolk, Virginia
  - Synergy Research Site, Richmond, Virginia
  - Synergy Research Site, Virginia Beach, Virginia
  - Synergy Research Site, Seattle, Washington
  - Synergy Research Site, Tacoma, Washington
  - Synergy Research Site, Wauwatosa, Wisconsin
- Canada (11):
  - Synergy Research Site, Kelowna, British Columbia
  - Synergy Research Site, Bridgewater, Nova Scotia
  - Synergy Research Site, Brampton, Ontario
  - Synergy Research Site, Cambridge, Ontario
  - Synergy Research Site, Greater Sudbury, Ontario
  - Synergy Research Site, London, Ontario
  - Synergy Research Site, Oshawa, Ontario
  - Synergy Research Site, Toronto, Ontario
  - Synergy Research Site, Mirabel, Quebec
  - Synergy Research Site, Pointe-Claire, Quebec
  - Synergy Research Site, Saint Romuald, Quebec

REFERENCES:
- [Derived] Cash BD, Sharma A, Walker A, Laitman AP, Chang L. Plecanatide for the treatment of chronic idiopathic constipation and irritable bowel syndrome with constipation: Post hoc analyses of placebo-controlled trials in adults with severe constipation. Neurogastroenterol Motil. 2023 Sep;35(9):e14632. doi: 10.1111/nmo.14632. Epub 2023 Jun 18. PMID 37332239
- [Derived] Rao SSC, Laitman AP, Miner PB Jr. Influence of Demographic Factors on Clinical Outcomes in Adults With Chronic Idiopathic Constipation Treated With Plecanatide. Clin Transl Gastroenterol. 2023 Jul 1;14(7):e00598. doi: 10.14309/ctg.0000000000000598. PMID 37162147
- [Derived] Moshiree B, Schoenfeld P, Franklin H, Rezaie A. The Effect of Acid Suppression Therapy on the Safety and Efficacy of Plecanatide: Analysis of Randomized Phase III Trials. Clin Ther. 2022 Jan;44(1):98-110.e1. doi: 10.1016/j.clinthera.2021.11.009. Epub 2022 Jan 25. PMID 35086735
- [Derived] Menees SB, Franklin H, Chey WD. Evaluation of Plecanatide for the Treatment of Chronic Idiopathic Constipation and Irritable Bowel Syndrome With Constipation in Patients 65 Years or Older. Clin Ther. 2020 Jul;42(7):1406-1414.e4. doi: 10.1016/j.clinthera.2020.05.012. Epub 2020 Jul 10. PMID 32660770
- [Derived] Miner PB Jr, Koltun WD, Wiener GJ, De La Portilla M, Prieto B, Shailubhai K, Layton MB, Barrow L, Magnus L, Griffin PH. A Randomized Phase III Clinical Trial of Plecanatide, a Uroguanylin Analog, in Patients With Chronic Idiopathic Constipation. Am J Gastroenterol. 2017 Apr;112(4):613-621. doi: 10.1038/ajg.2016.611. Epub 2017 Feb 7. PMID 28169285

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The data are correct and approved in the NDA. 1394 randomized subj.including 69 (index and non-index) duplicate subj. The index subj (21) were duplicate appeared the first time in the study and the same subject appeared in other studies or sites were non-index duplicate (48) who were excluded in the ITT population (1346).
Groups:
- Plecanatide 6 mg: Plecanatide tablets 6.0 mg QD for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Plecanatide 3.0 mg | Plecanatide 6 mg
Started | 452 | 453 | 441
Completed | 385 | 384 | 371
Not Completed | 67 | 69 | 70

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Plecanatide 3.0 mg | Plecanatide 6.0 mg | Total
Number analyzed (Participants) | 452 | 453 | 441 | 1346
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 46.4 [18 to 78] | 45.0 [18 to 79] | 45.1 [18 to 79] | 45.5 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 357 | 368 | 362 | 1087
  Male | 95 | 85 | 79 | 259

OUTCOME MEASURES:

1. Primary Outcome: Number of Durable Overall CSBM Responders , Mean Replacement Approach
Description: A durable overall CSBM responder was defined as a weekly CSBM responder for at least 9 of the 12 treatment weeks, included at least 3 of the last 4 weeks. A CSBM weekly responder was defined as a patient who has ≥ 3 Complete Spontaneous Bowel Movements (CSBMs) per week and an increase from baseline of ≥1 CSBM for that week. A CSBM was a bowel movement that occurred in the absence of laxative use within 24 hours and was associated with the feeling of complete evacuation.
Time Frame: 12-week Treatment Period
Population: The ITT (Intent-to-treat) population was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Plecanatide 3.0 mg | Plecanatide 6.0 mg
Number analyzed (Participants) | 452 | 453 | 441
Participants | 46 | 95 | 86

2. Secondary Outcome: Change From Baseline in CSBMs (CSBMS/Week) Over 12-week Treatment Period, Mean Replacement Approach
Description: A Complete Spontaneous Bowel Movement (CSBM) was a Bowel Movement (BM) that occurred in the absence of laxative use within 24 hours of the BM and the patient reported a feeling of complete evacuation. A weekly responder had 3 or more CSBMs and an increase of at least one CSBM from baseline in the same week.
Time Frame: 12-Week Treatment Period
Population: The ITT (Intent-to-treat) population was used for analysis.
Measure: Mean (Standard Deviation); unit: CSBMs per week
Arm/Group | Placebo | Plecanatide 3.0 mg | Plecanatide 6.0 mg
Number analyzed (Participants) | 452 | 453 | 441
CSBMs per week
  Baseline | 0.39 (0.570) | 0.32 (0.514) | 0.32 (0.509)
  Week 12 change from baseline | 1.45 (2.310) | 2.68 (3.891) | 2.39 (3.296)

3. Secondary Outcome: Change From Baseline in SBM (SBMs/Week) Over 12-week Treatment Period, Mean Replacement Approach
Description: The change from baseline in the number of Spontaneous Bowel Movement (SBM) over the 12-week Treatment Period was assessed. Baseline was the mean number of SBMs recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. The weekly SBM totals were derived from the daily diary entries reported during the Treatment Period in the BM and Symptom Diary.
Time Frame: 12-Week Treatment Period
Population: The ITT (Intent-to-treat) population was used for analysis.
Measure: Mean (Standard Deviation); unit: SBMs per week
Arm/Group | Placebo | Plecanatide 3.0 mg | Plecanatide 6.0 mg
Number analyzed (Participants) | 452 | 453 | 441
SBMs per week
  Baseline | 2.18 (2.032) | 1.97 (1.772) | 1.82 (1.824)
  Week 12 change from baseline | 1.37 (2.881) | 3.30 (4.628) | 3.24 (4.518)

4. Secondary Outcome: Change From Baseline in Stool Consistency Score Over the 12-week Treatment Period, Mean Replacement Approach
Description: The stool consistency of each bowel movement (BM) was assessed by patients using the 7-point Bristol Stool Form Scale [BSFS] from 1 to 7.
  1. = separate hard lumps like nuts (difficult to pass)
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on its surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges (passed easily)
  6. = fluffy pieces with ragged edges, a mushy stool
  7. = watery, no solid pieces (entirely liquid)
Time Frame: 12-Week Treatment Period
Population: The ITT (Intent-to-treat) population was used for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Plecanatide 3.0 mg | Plecanatide 6.0 mg
Number analyzed (Participants) | 452 | 453 | 441
score on a scale
  Baseline | 2.56 (1.114) | 2.52 (1.046) | 2.59 (1.171)
  Week 12 change from baseline | 0.83 (1.246) | 1.56 (1.504) | 1.47 (1.584)

5. Secondary Outcome: Change From Baseline in Straining Score Over 12-Week Treatment Period, Mean Replacement Approach
Description: Baseline was the mean of non-missing straining scores recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. The weekly average straining score was derived from the straining scores reported during the Treatment Period in the Daily Symptom Diary. The severity of straining during bowel movements was assessed on a 5-point Likert scale where 0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe.
Time Frame: 12-Week Treatment Period
Population: The ITT (Intent-to-treat) population was used for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Plecanatide 3.0 mg | Placebo | Plecanatide 6.0 mg
Number analyzed (Participants) | 453 | 452 | 441
score on a scale
  Baseline | 2.31 (0.835) | 2.30 (0.842) | 2.28 (0.894)
  Week 12 change from baseline | -0.70 (0.967) | -0.95 (1.027) | -1.00 (1.155)

ADVERSE EVENTS:
Description: The Intent-to-treat Safety (ITT-S) population (1389) was the enrolled population (1394) who received at least one dose of study drug.
Groups:
- Plecanatide 6.0 mg: Plecanatide tablets 3.0 mg QD for 12 weeks
Arm/Group | Placebo | Plecanatide 3.0 mg | Plecanatide 6.0 mg
Serious Adverse Events (participants affected / at risk) | 4/458 | 6/474 | 5/457
Other Adverse Events (participants affected / at risk) | 8/458 | 38/474 | 37/457
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=458) | Plecanatide 3.0 mg (N=474) | Plecanatide 6.0 mg (N=457)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=458) | Plecanatide 3.0 mg (N=474) | Plecanatide 6.0 mg (N=457)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 28 (28) | 26 (28)
Sinusitis (Infections and infestations) | 2 (2) | 10 (11) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes